CLINICAL TRIAL: NCT03743753
Title: Preoperative Education Intervention to Improve Patient Satisfaction and Optimize the Patient Experience in Breast Reconstruction: A Pilot, Feasibility Randomized Controlled Trial
Brief Title: Educational Session To Optimize Patient's Breast Reconstruction Experience at McMaster
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4844
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Breast Reconstruction; Patient Education
Keywords: Patient education; Satisfaction; Anxiety; Quality of life; Implant; Autologous; Breast reconstruction; Alloplastic
MeSH Terms: conditions — Personal Satisfaction; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The plastic surgeon will be blinded to participant's group allocation. The data analyst will also be blinded. They will be presented the data without group identification (i.e., Group A and Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive the current standard educational information from the surgeon along with an information package.
- Experimental (Experimental): The experimental group will receive an additional educational session before their operation about what to expect during their reconstructive journey, in addition to the current standard educational information from the surgeon along with an information package.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — The intervention is the educational session, which is a one-on-one session delivered by a research assistant using a visual aide on an iPad (power point presentation). The session is specifically tailored to the method of breast reconstruction (autologous or alloplastic) the patient will undergo and reviews the basics of their reconstruction, explains the normal in-hospital course and post-operative recovery, reviews potential complications and provides advice from previous breast reconstruction patients.
  Arms: Experimental

SUMMARY:
This pilot study uses a randomized controlled trial design to introduce an educational session for breast reconstruction patients. Participants will be randomly assigned to the (1) control group or the (2) experimental group. The control group will receive the current standard educational information from the surgeon along with an information package, while participants in the experimental group will also receive an additional education session before their operation about what to expect during their reconstructive journey. Satisfaction with care, anxiety about the procedure and recovery, and health related quality of life will be measured in all patients using established questionnaires. Additionally, feasibility outcomes will be reported and the results of this study will be used to demonstrate whether a larger version of this study can be successfully completed.

DETAILED DESCRIPTION:
This study is a feasibility, randomized controlled trial (RCT) to introduce a novel, pre-operative educational session for breast reconstruction patients. It will follow a single-center, 1:1 allocation, two-arm parallel group superiority design.

The primary objective of this trial is to determine feasibility of a larger, definitive RCT. The primary outcomes will allow for an accurate assessment of recruitment, study completion, efficient resource requirements and utilization, and treatment effect size. This will not only enhance the likelihood of success of a future RCT and allow us to foresee potential issues in study design, but also provide an opportunity for patient feedback on the educational intervention. The secondary objective is to address whether the novel, pre-operative educational intervention improves satisfaction (as measured with the BREAST-Q), health-related quality of life (as measured with the PROMIS-29) and decrease anxiety (as measured with the STAI for adults) in breast reconstruction patients at compared to the standard of care.

Participants will be randomly assigned to the (1) control group or the (2) experimental group. The control group will receive the current standard educational information from the surgeon along with an information package, while participants in the experimental group will also receive an additional education session before their operation.The session will be provided after the patient chooses their desired method of reconstruction and signs consent for their surgery. The session is specifically tailored to the method of breast reconstruction (autologous or alloplastic) the patient will undergo. It is a one-on-one session delivered by the research assistant using a visual aide on an iPad (power point presentation). The educational session reviews the basics of their reconstruction, explains the normal in-hospital course and post-operative recovery, reviews potential complications and provides advice from previous breast reconstruction patients. The information, visual aids, and lesson plan were created after a needs assessment of McMaster University breast reconstruction patients was performed (literature review, surgeon input, and semi-structured patient interviews).

The questionnaires (BREAST-Q, PROMIS-29 and STAI) will be administered to all participants at 4 time points: trial recruitment/initial consultation or preoperative appointment (1-2 weeks before surgery), and 3 follow-up time points (2-4 weeks, 3 months, and 6 months after surgery). If the participant is undergoing two-stage implant based reconstruction, the questionnaires will also be administered 1-2 weeks before the second surgery, and 2-4 weeks and 3 months after the second surgery. Qualitative interviews will be performed at 6 months post-operation with participants in the experimental group and control group. They will explore the patient perspective to identify ways to improve the content and delivery method of pre-operative education, and if in the control group, satisfaction with the standard care and information provided.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older
2. Able to understand and communicate in English
3. Patients who will be undergoing (or have had) a unilateral or bilateral mastectomy
4. Patients who will be undergoing primary breast reconstruction
5. Immediate or delayed breast reconstruction
6. Autologous (own tissue from the abdomen) or Alloplastic (tissue expander and implant) breast reconstruction.

Exclusion Criteria:

1. Breast conserving surgery (lumpectomy, partial mastectomy)
2. Reconstruction using only the latissimus dorsi muscle
3. Combined autologous and alloplastic reconstruction (e.g. latissimus dorsi and tissue expander)
4. Direct to implant reconstruction
5. Autologous reconstruction using tissue from a location other than the abdomen (e.g. buttock or thigh)
6. Seeking breast revision surgery or nipple reconstruction only
7. Patients who are unable to provide informed consent or are unable to complete quality of life questionnaires due to mental capacity or cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of the research study as measured by retention rate | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  The primary feasibility outcome will be retention rate at the 6 month-follow up. Retention rate is the percentage of enrolled participants who remain in the study until all study requirements are complete. A retention rate of >90% will indicate that a larger scale study is feasible.

SECONDARY OUTCOMES:
Patient Satisfaction | This questionnaire will be administered at the 1-2 week pre-operative visit and at the 2-4 weeks, 3 months and 6 months post-operation. (Also administered 1-2 weeks before, 2-4 weeks and 3 months after the 2nd surgery for implant based reconstruction).)
  This will be measured using the BREAST-Q questionnaire. The BREAST-Q is a patient reported outcome measure of patient satisfaction with breast reconstruction.The reconstructive module of the BREAST-Q will be administered. The questionnaire is composed of 10-13 sections depending on whether the participants underwent autologous or alloplastic reconstruction and whether the participant underwent radiation. All questions are answered on 3, 4, or 5 point Likert scales. The answers of each sections are totaled and compared to the equivalent Rasch transformed score. Zero represents the worst possible score and 100 represents the best.
Anxiety | This questionnaire will be administered at the 1-2 week pre-operative visit and at the 2-4 weeks, 3 months and 6 months post-operation. (Also administered 1-2 weeks before, 2-4 weeks and 3 months after the 2nd surgery for implant based reconstruction).)
  This will be measured using the Spielberger State-Trait Anxiety Inventory (STAI) for adults questionnaire. The STAI is a patient reported outcome that measures situational and trait anxiety. Of the two subscales, the State Anxiety Scale (S-Anxiety) evaluates the current state of anxiety. The Trait Anxiety Scale (T-Anxiety) evaluates relatively stable aspects of "anxiety proneness", including general states of calmness, confidence and security. The STAI has 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales. All items are rated on a 4-point Likert Scale. Scores range from 20 to 80, where higher scores indicate higher anxiety.
Health-related quality of life | This questionnaire will be administered at the 1-2 week pre-operative visit and at the 2-4 weeks, 3 months and 6 months post-operation. (Also administered 1-2 weeks before, 2-4 weeks and 3 months after the 2nd surgery for implant based reconstruction).)
  This will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS-29) questionnaire. The PROMIS-29 is a generic health-related quality of life survey that assesses 7 domains (physical function, pain interference, fatigue, sleep disturbance, anxiety, depression, satisfaction with participation in social roles) and is designed to measure self-reported physical, mental and social health and wellbeing. The questions are answered on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. In symptom-oriented domains (pain interference, fatigue, sleep disturbance, anxiety and depression) higher scores represent worse symptomatology. In function-oriented domains (physical functioning and social role) higher scores represent better functioning.
Feasibility measure: Recruitment rate | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is recruitment rate, the number of participants who were enrolled in the study out of the number who were assessed for eligibility, as described as a percentage. A recruitment rate of >70% will indicate that a larger scale study is feasible.
Feasibility measure: Compliance rate | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is compliance rate, the percentage of participants who were randomized to the experimental group who completed the intervention.
Feasibility measure: Percent of patients who meet eligibility criteria | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is eligibility, the percentage of patients who were assessed for eligibility who meet all the eligibility criteria. An eligibility percentage of >80% will indicate that a larger scale study is feasible.
Feasibility measure: Time assessment | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is a time assessment, the number of months it take to complete the research study.
Feasibility measure: Budget assessment | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is a budget assessment, the amount of money and the allocation of money that is required to complete the study. This will be compared to the budget designed prior to study commencement.
Feasibility measure: Personnel time | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is personnel time, the number of hours and the allocation of hours each member of the research time has dedicated to completing this study.
Feasibility measure: Treatment effect size and variance of the primary, secondary outcome. | This will be calculated through study completion, an average of 1 year, at the time when every enrolled participant is set to complete the final follow up.
  This secondary, feasibility outcome is treatment effect size. This will be calculated using the mean difference between the control and experimental groups of the Satisfaction with Information subscale in the BREAST-Q at the 3 month follow up time. The mean difference will be divided by the pooled standard deviation (variance) to determine the effect size.

CONTACTS AND LOCATIONS:
Overall Officials: Sophocles Voineskos, MD, MSc., Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario